CLINICAL TRIAL: NCT06049849
Title: Can Participants With Chronic Stroke Regain Living Independence by Daily Energizing With a Biophoton Generator
Brief Title: Can Patients With Chronic Stroke Regain Living Independence by Daily Energizing With Biophoton Generators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Institute of All Medicines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022/09/27
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Stroke
Keywords: stroke, paralysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study is a randomized, triple-blinded, placebo-controlled prospective intervention clinical research. All patients with chronic stroke will participate in the live-in observational study by sleeping on Tesla MedBed in a special hotel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All products are individual coded. All other visible characters are identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental): Active Biophoton Generators are placed under the hotel bed.
  Interventions: Device: Biophoton Energizing Brain and Whole Body
- Control Group (Placebo Comparator): Placebo-products are placed under the hotel bed.
  Interventions: Device: Biophoton Energizing Brain and Whole Body

INTERVENTIONS:
Device: Biophoton Energizing Brain and Whole Body — The patient is to be energized within a strong biophoton field which is constantly generated by active biophoton generators.

SUMMARY:
Study objective The purpose of this clinical research is to verify if the patient with chronic stroke can regain the ability of living independently after daily using Testa BioHealing® Biophoton Generators to increase the energy of the brain and other parts of the body.

Study design This study is a randomized, triple-blinded, placebo-controlled prospective intervention clinical research. At least 46 patients with chronic stroke will participate in the live-in observational study in a Tesla MedBed Center.

Study patient population The adult patient with a chronic stroke which was defined as a stroke occurred at least 6 months ago with a significant disability unable to have an independent life, is to be considered as a qualified participant.

DETAILED DESCRIPTION:
Investigational product and mode of administration The hotel bed is powered by a standardized set of 14 biophoton generators of 32-Oz size, which was previously tested as safe and effective. The active device is FDA registered over-the-counter (OTC) medical device. The device can be used by anyone who wants to increase blood circulation and reduce bodily pains, according to the label claims. For this study, the active or inactive devices will be labeled with individual codes. The participant, caregiver and the study staff cannot know if the hotel room is equipped with a set of active or inactive devices. When the participant is lying on the hotel bed, she/he may or may not receive biophotons. The study physician, participant or the caregiver will record the ADL and other changes, and answer the standard study questionnaires at the baseline, 2, or 4 weeks after study treatment, respectively.

Study procedure Each of all participants assigned to the Control or Treatment Group will be continually treated with the current standard of care (SOC), if any. The Control group will use the coded placebo devices, and the Treatment Group will use the coded treatment product. All coded products will be packed with the same container with the same size and weight. Each participant will use the Treatment or Control device at least for 8-hours every day for 4-weeks during sleep and any daytime during the day. Each participant and caregiver will be guided by the study physician to use Katz Index of Independence in Activities of Daily Living (ADL) to measure the level of life independence. The study physician will perform neurological examination. Stroke Impact Scale (SIS) for stroke-specific health status measurement, SF-36 questionnaires (SF-36) to measure life quality, Electroencephalography (EEG) test, and Bio-Well energy test, will be conducted respectively at the baseline, 2 or 4 weeks after the study treatment. SIS and SF-36 questionnaires will be recalled 4 weeks before the baseline for each participant.

Comparator and mode of administration The same shape, size, and weight of the device without generating biophoton is to be labelled with individual codes and used as a comparator. The comparator device will be placed in the same way as the Treatment device in the hotel room during the designed study period.

Study duration Estimated date of the first participant enrolled: May 2023. The estimated date of the last patient completed: December 2023. The participants randomized in the Control group will be switched to the Treatment after observing the placebo effects for four weeks. They will be treated with the active device for 4-weeks for self-comparison analysis.

Duration of treatment Participants in the Control and Treatment Groups will actively participate in the study for 4-weeks. Each participant and caregiver will answer the standard study questionnaires at the baseline, 2 or 4 weeks of the study, respectively. The participants randomized in the Control will participate in the study for a total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18-years or older and can live in a hotel
* Must have a caregiver willing to support the participant's full involvement in the study and can assist to complete all study questionnaires
* Can provide informed consent (maybe assisted by Caregiver)
* Has evidence of a clinical diagnosis of stroke occurred at least 6 months ago.
* Has a disability unable to be living independently per Caregiver
* Can complete all study procedures during the study
* Must be fluent in English (or the Caregiver can fully translate)

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by the Caregiver or by the clinical study medical professional
* Who relies on ventilators
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include severe chronic pulmonary disease, history of uncontrolled seizures, acute or chronic infectious illness, kidney failure, etc.
* Is participating in another investigational drug or device trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Regain Life Independence by Normalizing Activities of Daily Living (ADL). | 0-2 weeks, 0-4 weeks after starting the study treatment.
  If the damaged brain is repaired, the participant can perform daily activities.

SECONDARY OUTCOMES:
Neurologic Examination Using a Standard Neurologic Exam Form to Measure Neurologic Function | 0-2 weeks, 0-4 weeks after starting the study treatment.
  The study physician will conduct the standardized neurologic examinations
Stroke Impact Scale (SIS) to Reflect Paralysis Status Change (fully recovery =300) | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Under study physician's guidance, participant will answer the standard questionnaires.
Brain injury status detected with EEG (electroencephalogram). | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Brain injury exists at the baseline and can be repaired with biophotons.
Life Quality Improvement Measured with a Standard SF-36 Questionnaire | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Using Short Form Health Survey (SF-36) to measure life quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Tesla MedBed Center at Butler-PA, Butler, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All individual participants' identification information will be kept confidential. All data report forms will have the subject number. The study report and scientific publication will not show any identifiable information of the patient.